CLINICAL TRIAL: NCT06350149
Title: A Pilot and Feasibility Study to Evaluate High vs Low Glycemic Index Mixed Meal Tolerance Test in Adolescents and Young Adults With Cystic Fibrosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Tanicia Daley, Professor, Emory University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: STUDY00004637; 1R21DK128731-01A1 (NIH)
Record Dates: First submitted 2024-03-28; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Glycemic Index; Cystic Fibrosis Related Diabetes
MeSH Terms: conditions — Cystic Fibrosis | interventions — Sugar-Sweetened Beverages

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SSB+ HI- GI (Experimental): All standardized mixed meal challenges will be similar in calories (kcal) and percent of calories from carbohydrates (45%), protein (15%), and fat (40%). Each meal will provide 1/3rd of the subject's estimated kcal needs per current CF nutrition guidelines
  Interventions: Other: Sugar Sweetened Beverages (SSB); Other: Hi GI
- SSB + LO- GI (Experimental): All standardized mixed meal challenges will be similar in calories (kcal) and percent of calories from carbohydrates (45%), protein (15%), and fat (40%). Each meal will provide 1/3rd of the subject's estimated kcal needs per current CF nutrition guidelines
  Interventions: Other: Sugar Sweetened Beverages (SSB); Other: Lo GI
- NSSB+ HI- GI (Experimental): All standardized mixed meal challenges will be similar in calories (kcal) and percent of calories from carbohydrates (45%), protein (15%), and fat (40%). Each meal will provide 1/3rd of the subject's estimated kcal needs per current CF nutrition guidelines
  Interventions: Other: Hi GI
- NSSB+ LO- GI (Experimental): All standardized mixed meal challenges will be similar in calories (kcal) and percent of calories from carbohydrates (45%), protein (15%), and fat (40%). Each meal will provide 1/3rd of the subject's estimated kcal needs per current CF nutrition guidelines
  Interventions: Other: Lo GI

INTERVENTIONS:
Other: Sugar Sweetened Beverages (SSB) — The following are considered SSBs: non-diet soft drinks/sodas, flavored juice drinks, sweetened tea, energy drinks, and electrolyte replacement drinks.
  Arms: SSB + LO- GI; SSB+ HI- GI
Other: Hi GI — The Glycemic Index of the high-GI meals will be at least 75
  Other Names: Hight Glycemic Index Meal
  Arms: NSSB+ HI- GI; SSB+ HI- GI
Other: Lo GI — The Glycemic Index of the low- -GI meals will not be higher than 55.
  Other Names: Low Glycemic Index Meal
  Arms: NSSB+ LO- GI; SSB + LO- GI

SUMMARY:
The goal of this study is to determine the extent to which excess dietary simple sugars serve as a secondary mediating factor in Cystic fibrosis-related diabetes (CFRD) development. The main questions it aims to answer are:

* Whether conducting a randomized 2x2 factorial design that evaluates acute postprandial changes in glucose over 2 hours following ingestion of a mixed meal challenge that varies by glycemic index and consumption of a sugar-sweetened beverage is acceptable and feasible.
* What are the preliminary changes in postprandial hyperglycemia, islet cell function, and incretin response to a high or low Glycemic Index mixed meal tolerance test (MMTT) with and without Sugar-Sweetened Beverages (SSB) in adolescents and young adults with CF

Participants will be randomized to a mixed diet and blood will be drawn before and after the mixed meal challenge.

DETAILED DESCRIPTION:
Cystic fibrosis-related diabetes (CFRD) is one of the most common co-morbidities seen in CF and significantly increases morbidity and mortality. The prevalence of CFRD increases with age with approximately 20% of adolescents and 50% of adults in the 3rd and 4th decade of life carrying the diagnosis. Although a diagnosis of CFRD is uncommon in children less than 10 years of age, research studies show that abnormal glucose tolerance is found in about 40% of CF toddlers and school-age children. Mechanisms leading to the development of CFRD are incompletely understood. For several years, the predominant theory of pancreatic endocrine dysfunction was based on the theory of "collateral damage" which results in impairment of β-cell function due to loss of islet cells. In addition to experiencing reduced beta cell mass, individuals with CF have a diminished incretin effect that contributes to impaired insulin secretion. Postprandial hyperglycemia is not uncommon for individuals with CF irrespective of their glucose tolerance and during an OGTT failure to suppress glucagon results in hyperglycemia. Unfortunately, mechanisms involved in dysregulated glucagon release and its contribution to hyperglycemia in CF are poorly understood.

The CF diet is typically high in energy-dense, nutrient-poor foods. Individuals with CF require high-energy, high-fat diets to maintain their hypermetabolic state and offset malabsorption, with current CF dietary guidelines recommending an energy intake of 1.2 to 1.5 times that of the general population. To date, there is a paucity of studies that rigorously investigate the metabolic sequelae that high GI foods and SSB have on the metabolic profile of individuals with CF. The study team proposes that a diet high is SSBs and high GI foods induces more oxidative stress due to postprandial hyperglycemia, impairs insulin secretion, and exacerbates glucose abnormalities in CF.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Diagnosis of CF based on the presence of two known CF causing mutations and/or positive sweat test
* Pancreatic insufficiency
* Baseline dietary consumption of >10% total kcal from added sugars and self-reported consumption of >/= sugar-sweetened beverages per week

Exclusion Criteria:

* Current use or anticipated use of medication that is known to raise or lower blood glucose in the past 4 weeks.
* Oral or IV glucocorticoid current or previous use in the past 4 weeks will prohibit enrollment in the study.
* Recent pulmonary exacerbation within 3 weeks of enrollment and/or an acute illness requiring a change in antibiotics will also exclude participants.
* BMI below the 5th percentile or greater than the 95th percentile for age and sex
* FEV1 <40% or awaiting a lung transplant;
* Prior lung or liver transplant or kidney or liver dysfunction.
* Use of CFTR modulators is not an exclusion criterion. Rather, for patients recently started on CFTR modulators, we will wait to enroll in the study until on CFTR modulator for at least 2 months.
* Diagnosis of CF liver disease.
* Uncontrolled exocrine pancreatic insufficiency/malabsorption
* Diagnosis of CFRD
* G-tube feeds (bolus and/or continuous)
* Current enrollment in another intervention study
* Changes in diet to lose or gain weight
* Gluten allergy or intolerance
* Current pregnancy or lactation or plans to become pregnant during study period
* History of drug or alcohol abuse
* Restrictive dietary patterns (e.g, vegan, ketogenic, intermittent fasting) for more than one month within the last two months prior to screening.
* More than 5% body weight change within 2 months of screening visit or Day 1 of mixed meal tolerance test

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | 2 years
  Recruitment rate of participants. Goal is to recruit 3 participants per month.
Refusal Rate | 2 years
  Refusal rates for participation. 20%of screened participants will refuse to participate
Investigator Fidelity | 2 years
  Capacity of the research team to manage the intervention. Goal is >85%.
Participant Fidelity | 2 years
  Feasibility of data collection, including primary and secondary outcome measures. Goal is >85%
Acceptability | 2 years
  Acceptability and burden of intervention on participants. Likert scale response of >3(out of 5) on post study evaluation that study is not burdensome and acceptable
Retention Rates | 2 years
  Retention rates as the participants complete the intervention. Goal is >80%
Recruitment | 2 years
  Length of time it takes to recruit enough participants into the study. Goal is to recruit all patients by the end of second quater of the second year.

SECONDARY OUTCOMES:
Change in plasma Cysteine (Cys) | Baseline, 2 hours
  Systemic redox balance will be assessed by high performance liquid chromatography measurement of plasma CyS
Change in plasma Cystine (CySS) | Baseline, 2 hours
  Systemic redox balance will be assessed by high performance liquid chromatography measurement of plasma CySS
Change in plasma Glutathione (GSH) | Baseline, 2 hours
  Systemic redox balance will be assessed by high performance liquid chromatography measurement of plasma GSH
Change in plasma Glutathione Disulfide (GSSG) | Baseline, 2 hours
  Systemic redox balance will be assessed by high performance liquid chromatography measurement of plasma GSSG
Change in redox potentials (EhCys/ CySS and EhGSH/GSSG) | Baseline, 2 hours
  Systemic redox balance will be assessed by high performance liquid chromatography measurement of plasma redox potentials (EhCys/CySS and EhGSH/GSSG)
Insulinogenic index | Baseline, 30 mins
  It estimates the efficiency of glucose disposal in the early phase of stimulated insulin secretion.
Whole body insulin sensitivity index (WBISI-Matsuda) | 2 hours
  Whole-body insulin sensitivity (WBISI) will be assessed by the method of Matsuda and Defronzo, which combines both hepatic and peripheral tissue insulin sensitivity. HOMA-IR will provide a reflection of hepatic insulin resistance.
Disposition Index | 2 hours
  The disposition index, a measure of beta cell function for a given level of insulin resistance, will be calculated as: (WBISI) × (insulin secretion)
Change in plasma Eh Cys/CySS | Baseline, 2 hours
  Systemic redox balance will be assessed by high performance liquid chromatography measurement of plasma redox potentials EhCys/CySS
Change in incremental glucose AUC | Baseline, 120 minutes
  AUC: area under the curve from baseline to 120 minutes
Changes in Plasma insulin | Baseline, 2 hours
  Changes in post prandial plasma insulin levels will be measured.
Changes in Plasma C-peptide | Baseline, 2 hours
  Changes in post prandial plasma C-peptide levels will be measured.
Changes in Plasma Glucagon | Baseline, 2 hours
  Changes in post prandial plasma glucagon levels will be measured.
Changes in Plasma Incretins: glucagon-like peptide-1 (GLP-1) | Baseline, 2 hours
  Blood for determination of active glucagon-like peptide-1 (GLP-1) will be collected until the 30-minute timepoint in tubes filled with protease inhibitors. GLP-1 will be measured in duplicate by ELISA . The total and iAUC30 will be determined
Changes in Plasma Incretins: total glucose-dependent insulinotropic polypeptide (GIP) | Baseline, 2 hours
  Blood for determination of GIP will be collected until the 30-minute timepoint in tubes filled with protease inhibitors. GLP-1 will be measured in duplicate by ELISA . The total and iAUC30 will be determined

CONTACTS AND LOCATIONS:
Overall Officials: Tanicia Daley, MD, MPH, Principal Investigator — Emory University
Locations (1):
- Center for Advanced Pediatrics: Emory Healthcare, Atlanta, Georgia, United States